CLINICAL TRIAL: NCT06459687
Title: Efficacy and Safety of Socazolimab Combined With Chemotherapy With or Without Bevacizumab as First-Line Treatment in Persistent, Recurrent, or Metastatic Cervical Cancer: A Randomized, Double-blind, Placebo-controlled Phase III Study
Brief Title: Phase III Study of Socazolimab as First-Line Treatment in Persistent, Recurrent, or Metastatic Cervical Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKAB001-LEES-2024-01
Record Dates: First submitted 2024-06-03; First posted 2024-06-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socazolimab+Chemotherapy±Bevacizumab (Experimental): 6~8 cycles of Socazolimab (5 mg/kg) + cisplatin (50 mg/m2) /carboplatin (AUC5) + paclitaxel (175 mg/m2) ± Bevacizumab (15 mg/kg), Q3w.
  Followed with Socazolimab (5 mg/kg), Q3w.
  Interventions: Drug: Socazolimab+cisplatin/carboplatin+paclitaxel+Bevacizumab
- Placebo+Chemotherapy±Bevacizumab (Placebo Comparator): 6~8 cycles of placebo (5 mg/kg) + cisplatin (50 mg/m2) /carboplatin (AUC5) + paclitaxel (175 mg/m2) ± Bevacizumab (15 mg/kg), Q3w.
  Followed with placebo (5 mg/kg), Q3w.
  Interventions: Drug: Placebo+cisplatin/carboplatin+paclitaxel+Bevacizumab

INTERVENTIONS:
Drug: Socazolimab+cisplatin/carboplatin+paclitaxel+Bevacizumab — 6~8 cycles of Socazolimab (5 mg/kg) + cisplatin (50 mg/m2) /carboplatin (AUC5) + paclitaxel (175 mg/m2) ± Bevacizumab (15 mg/kg), Q3w.
  Followed with Socazolimab (5 mg/kg), Q3w.
  Arms: Socazolimab+Chemotherapy±Bevacizumab
Drug: Placebo+cisplatin/carboplatin+paclitaxel+Bevacizumab — 6~8 cycles of placebo (5 mg/kg) + cisplatin (50 mg/m2) /carboplatin (AUC5) + paclitaxel (175 mg/m2) ± Bevacizumab (15 mg/kg), Q3w.
  Followed with placebo (5 mg/kg), Q3w.
  Arms: Placebo+Chemotherapy±Bevacizumab

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Socazolimab combined with chemotherapy with or without bevacizumab as first-Line treatment in persistent, recurrent, or metastatic cervical cancer. The main question it aims to answer is:

Does Socazolimab combined with chemotherapy with or without bevacizumab better benefit patients with persistent, recurrent, or metastatic cervical cancer as first-line treatment compared with placebo combined with chemotherapy with or without bevacizumab.

Participants will be treated with Socazolimab/placebo + chemotherapy ± bevacizumab) for 6~8 cycles (Q3w), following maintenance treatment of Socazolimab/placebo (Q3w).

ELIGIBILITY:
Inclusion Criteria:

* 1. Able to understand and voluntarily signed written informed consent. Informed consent must be signed prior to specified study procedure.
* 2. Age ≥ 18 years and ≤75 years on the date of signing the informed consent, female.
* 3. ECOG Physical fitness score was 0 or 1.
* 4. Life expectancy ≥ 3 months.
* 5. Histologically confirmed cervical cancer that cannot be cured by surgery or radiotherapy/concurrent chemoradiotherapy.
* 6. Have at least one measurable tumor lesion examined by CT or MRI according to RECIST v1.1 criteria;
* 7. All subjects must provide archived or freshly obtained tumor tissue samples (formalin-fixed paraffin-embedded [FFPE] tissue wax blocks or at least 5 unstained tumor tissue section samples, preferably newly obtained tumor tissue samples) within the previous 5 years of randomization.
* 8. Laboratory examination results during the screening period indicate that the subject has good organ function.
* 9. Effective contraception should be used by fertile female subjects from the signing of informed consent until 180 days after the last administration of the study drug.

Exclusion Criteria:

* 1. Other histopathological types of cervical cancer, such as small cell carcinoma, clear cell carcinoma, sarcoma, etc.
* 2. Prior anti-angiogenic therapy (e.g., bevacizumab), immune checkpoint inhibitors (e.g., anti-PD-1 antibody, anti-PD-L1 antibody, anti-CTLA-4 antibody, etc.), or targeting immune costimulators (e.g. antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.) and any treatment targeting the immune mechanism of tumor.
* 3. Active or potentially recurring autoimmune disease.
* 4. Patients with other active malignant tumors within 3 years prior to randomization.
* 5. Participants who had participated in other clinical studies and used other clinical trial drugs within 4 weeks before randomization.
* 6. Major surgery, open biopsy or significant trauma within 4 weeks before randomization; Or an expected major surgical treatment during the study.
* 7. Anti-tumor therapy within 4 weeks before randomization.
* 8. Severe infection occurring within 4 weeks prior to randomization.
* 9. Vaccination within 4 weeks prior to randomization.
* 10. Received immune-modulating drugs (such as thymosin, interferon, interleukin-2) within 2 weeks before randomization.
* 11. Use of systemic antibacterial, antiviral, or antifungal drugs within 2 weeks prior to randomization.
* 12. Subjects requiring systemic treatment with corticosteroids (> 10 mg/ day of prednisone or equivalent doses of corticosteroids) or other immunosuppressive drugs within 2 weeks prior to randomization.
* 13. Clinically significant hydronephrosis that cannot be relieved by nephrostomy or ureteral stenting as determined by the investigator.
* 14. Central nervous system metastatic or cancerous meningitis.
* 15. Uncontrolled pleural, pericardial, or peritoneal effusions requiring repeated drainage (more frequently than monthly).
* 16. Known primary or secondary immunodeficiency, including a positive test for human immunodeficiency virus (HIV) antibodies.
* 17. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* 18. Known active tuberculosis; Known active treponema pallidum infection.
* 19. known history of severe hypersensitivity to other monoclonal antibodies.
* 20. Known contraindications to cisplatin/carboplatin, paclitaxel, or allergies to any components.
* 21. Previous and/or current presence of interstitial lung disease, pneumoconiosis, drug-related pneumonia, severe impairment of pulmonary function, etc., that may interfere with the detection and management of suspected drug-related pulmonary toxicity.
* 22. Subjects with active viral hepatitis B, inactive or asymptomatic carriers of hepatitis B virus (HBV) (positive for hepatitis B surface antigen [HBsAg]) with HBV DNA > 500 IU/mL or > 2500 copies/mL), and subjects with active viral hepatitis C.
* 23. Active or documented inflammatory bowel disease.
* 24. Any of the following cardiovascular diseases: a) myocardial infarction, unstable angina pectoris, pulmonary embolism, aortic dissection, deep vein thrombosis, and any arterial thromboembolism event occurred within 6 months before randomization; b) New York Heart Association (NYHA) heart function grade ≥ II heart failure; c) There is a serious arrhythmia that requires drug intervention; Patients with asymptomatic atrial fibrillation with stable ventricular rate were admitted; d)Left ventricular ejection fraction (LVEF) < 50%.
* 25. NCI CTCAE v5.0 ≥ 2 grade peripheral neuropathy.
* 26. Not recovered from toxicity of previous antitumor therapy.
* 27. Pregnant or lactating women.
* 28. Any condition (such as another serious illness or psychiatric disorder) that the investigator believes may result in a risk for acceptance of the study drug or that would interfere with the evaluation of the study drug or with the safety of the subjects or the interpretation of the study results.
* 29. Known contraindications to bevacizumab or allergies to any of its components, or the presence of any medical conditions that could affect the safety of bevacizumab administration.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization to date of death from any cause, assessed up to 100 months.

SECONDARY OUTCOMES:
PFS (assessed by BICR, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
ORR (assessed by BICR, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
DoR (assessed by BICR, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
DCR (assessed by BICR, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
TTR (assessed by BICR, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
PFS (assessed by investigators, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
ORR (assessed by investigators, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
DoR (assessed by investigators, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
DCR (assessed by investigators, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
TTR (assessed by investigators, based on RECIST v1.1) | From date of randomization to date of death from any cause or lost of visit, whichever came first, assessed up to 100 months.
Safety: adverse events, clinical abnormalties | from written informed concent to 90 days after last dose
Tmax | from 30min before first dose to 30 days after last dose
Cmax | from 30min before first dose to 30 days after last dose
T1/2 | from 30min before first dose to 30 days after last dose
Immunogenicity | from 30min before first dose to 30 days after last dose
  ADA, NAb
Health-related quality of life (HRQoL) | from screening to end of treatment visit, up to 100 months
  using EORTC QLQ-C30 Questionnaire
PD-L1 status | up to 100 months

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang